CLINICAL TRIAL: NCT03796169
Title: Effect of Intervention for Improving Colonoscopy Quality is Associated With the Personal Characteristics of the Endoscopist
Brief Title: Effect of Intervention for Colonoscopy Quality is Associated With the Personal Characteristics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Saint Vincent's Hospital, Korea (Other); Uijeongbu St. Mary Hospital (Other)
Responsible Party: Principal Investigator, Bo-In Lee, Professor, MD, PhD, Seoul St. Mary's Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: XC15FIMI0020K
Record Dates: First submitted 2018-12-16; First posted 2019-01-08 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Colonoscopy; Human Characteristics
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopist (Experimental): Intervention for personal notification, open notification and colonoscopy quality education by a GI faculty
  Interventions: Behavioral: Personal notification; Behavioral: Open notification; Behavioral: Education

INTERVENTIONS:
Behavioral: Personal notification — Baseline quality indicators of each endoscopist were measured and those were notified individually.
Behavioral: Open notification — Quality indicators were measured for 3 months after 1st interventions and those were notified openly
Behavioral: Education — Quality indicators were measured for 3 months after 2nd interventions and educated the importance of colonoscopy quality by a GI faculty

SUMMARY:
This study aims to investigate whether the personal characteristics of the endoscopist is associated with effect of interventions for colonoscopy quality improvement.

This is a prospective, 9-month, multicenter, single-blind study. Baseline quality indicators including adenoma detection rate, polyp detection rate, withdrawal time and adenomas per colonoscopy of each endoscopist were measured in the health promotion centers of academic hospitals for 3 months. Follow-up measurements of quality indicators were repeated every 3 months after each interventions (personal notification of quality indicators, open notification of quality indicators, and colonoscopy quality education by a GI faculty. At the end of the study, personal characteristics of each endoscopist was evaluated using fear of negative evaluation scale, cognitive flexibility inventory, and almost perfect scale.

DETAILED DESCRIPTION:
Suboptimal colonoscopy quality is associated with development of interval colorectal cancer and colorectal cancer-related death. It is uncertain how to improve colonoscopy quality effectively. The quality of screening colonoscopy for colorectal cancer depends on the endoscopist who performed the examination. The aim of this study was to investigate the impact of endoscopists' personal characteristics on the quality of colonoscopy and effectiveness of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Highly experienced board-certified gastroenterologists performed colonoscopies in health screening endoscopy centers.
* Endoscopists who sign the consent
* Patients for quality indicators of endoscopists

  * routinely perform outpatient screening, surveillance and diagnostic colonoscopy (first-time screening colonoscopies performed and had no previous colonoscopy within 3 years).

Exclusion Criteria:

* endoscopists who refuse to sign the consent
* Patients for quality indicators of endoscopists

  * Known hereditary polyposis syndrome, Inflammatory bowel disease, those with surgically altered anatomy, undergone previous colonoscopy within 3 years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Measurement of overall adenoma detection rate | 9 months
  Primary outcome measures include overall adenoma detection rate.
Measurement of adenoma detection rate after personal notification | 3 months after personal notification
  Primary outcome measures include adenoma detection rate after personal notification
Measurement of adenoma detection rate after open notification | 3 months after open notification
  Primary outcome measures include adenoma detection rate after open notification
Measurement of adenoma detection rate after education | 3 months after education
  Primary outcome measures include adenoma detection rate after education

SECONDARY OUTCOMES:
Measurement of overall polyp detection rate | 9 months
  Secondary outcome measures include overall polyp detection rate.
Measurement of overall withdrawal time | 9 months
  Secondary outcome measures include overall withdrawal time.
Measurement of overall adenomas per colonoscopy | 9 months
  Secondary outcome measures include overall adenomas per colonoscopy.
Measurement of polyp detection rate after personal notification | 3 months after personal notification
  Primary outcome measures include polyp detection rate after personal notification
Measurement of polyp detection rate after open notification | 3 months after open notification
  Primary outcome measures include polyp detection rate after open notification
Measurement of polyp detection rate after education | 3 months after education
  Primary outcome measures include polyp detection rate after education
Measurement of withdrawal time after personal notification | 3 months after personal notification
  Primary outcome measures include withdrawal time after personal notification
Measurement of withdrawal time after open notification | 3 months after open notification
  Primary outcome measures include withdrawal time after open notification
Measurement of withdrawal time after education | 3 months after education
  Primary outcome measures include withdrawal time after education
Measurement of adenomas per colonoscopy after personal notification | 3 months after personal notification
  Primary outcome measures include adenomas per colonoscopy after personal notification.
Measurement of adenomas per colonoscopy after open notification | 3 months after open notification
  Primary outcome measures include adenomas per colonoscopy after open notification
Measurement of adenomas per colonoscopy after education | 3 months after education
  Primary outcome measures include adenoma detection rate after education

CONTACTS AND LOCATIONS:
Overall Officials: Bo-In Lee, MD, PhD, Principal Investigator — Division of Gastroenterology; Seoul St. Mary's hospital
Locations (1):
- Division of Gastroenterology; Seoul St. Mary's hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coe SG, Crook JE, Diehl NN, Wallace MB. An endoscopic quality improvement program improves detection of colorectal adenomas. Am J Gastroenterol. 2013 Feb;108(2):219-26; quiz 227. doi: 10.1038/ajg.2012.417. Epub 2013 Jan 8. PMID 23295274
- [Background] Shaukat A, Oancea C, Bond JH, Church TR, Allen JI. Variation in detection of adenomas and polyps by colonoscopy and change over time with a performance improvement program. Clin Gastroenterol Hepatol. 2009 Dec;7(12):1335-40. doi: 10.1016/j.cgh.2009.07.027. Epub 2009 Aug 7. PMID 19665583
- [Background] Jover R, Zapater P, Bujanda L, Hernandez V, Cubiella J, Pellise M, Ponce M, Ono A, Lanas A, Seoane A, Marin-Gabriel JC, Chaparro M, Cacho G, Herreros-de-Tejada A, Fernandez-Diez S, Peris A, Nicolas-Perez D, Murcia O, Castells A, Quintero E; COLONPREV Study Investigators. Endoscopist characteristics that influence the quality of colonoscopy. Endoscopy. 2016 Mar;48(3):241-7. doi: 10.1055/s-0042-100185. Epub 2016 Feb 4. PMID 26845473
- [Derived] Choi HH, Sung SY, Lee BI, Cho H, Jung Y, Park JM, Cho YS, Lee KM, Kim SW, Choi H, Chae HS, Choi MG. The Effect of Intervention for Improving Colonoscopy Quality Is Associated with the Personality Traits of Endoscopists. Gut Liver. 2024 Mar 15;18(2):265-274. doi: 10.5009/gnl220280. Epub 2023 May 9. PMID 37158042